CLINICAL TRIAL: NCT01754402
Title: A Phase I-II Study of the Combination of Bendamustine and Pomalidomide With Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Bendamustine + Pomalidomide + Dex in R/R Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cristina Gasparetto (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Cristina Gasparetto, Sponsor Investigator, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00040206; PO-MM-PI-0045 (Other: Celgene)
Record Dates: First submitted 2012-11-27; First posted 2012-12-21 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Dose escalation with 3+3 cohort design plus Dose expansion at the Maximum tolerated dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: benda 120mg + pom 3mg (Experimental): * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  Interventions: Drug: Bendamustine; Drug: Pomalidomide; Drug: Dexamethasone
- Cohort 2: benda 120mg + pom 4mg (Experimental): * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  Interventions: Drug: Bendamustine; Drug: Pomalidomide; Drug: Dexamethasone
- Expansion (Experimental): * Pomalidomide 3mg: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine 120 mg: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  Interventions: Drug: Bendamustine; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered intravenously over 1 hour (if using Treanda) or over 10 minutes (if using Bendeka) on day 1, every 28 days for 12 cycles.
  Other Names: Treanda; Bendeka
Drug: Pomalidomide — Pomalidomide will be administered once daily orally (PO) on days 1-21, every 28 days until disease progression or death.
  Other Names: CC-4047; Pomalyst
Drug: Dexamethasone — Dexamethasone will be administered weekly orally or intravenously on days 1, 8, 15, and 22 every 28 days until disease progression or death. After 6 cycles of treatment, the dose may be reduced to 20mg at investigator's discretion. For subjects ≥ 75 years of age, the starting dose of dexamethasone is 20 mg/day on Days 1, 8, 15 and 22 of each 28-day treatment cycle.

SUMMARY:
This study is designed as a phase I-II, open label, dose finding study.

Study treatment will be as follows, in 28 day cycles:

* Pomalidomide: once daily orally (PO) dosing on days 1-21, every 28 days
* Bendamustine: once intravenously (IV) dosing on day 1, every 28 days
* Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22.

After completing 6 cycles of treatment, dexamethasone may be decreased to 20mg per investigator discretion. After completing 12 cycles of treatment, patients will proceed to the maintenance phase of the study. Patients will receive Pomalidomide on day 1-21, every 28 days and dexamethasone on days 1, 8, 15, and 22 every 28 days until time of progression.

DETAILED DESCRIPTION:
PRIMARY ENDPOINTS:

Phase I • Determination of the MTD of the combination therapy

Phase II:

• Response rate (CR+PR)

SECONDARY ENDPOINTS:

* Overall Response Rate (ORR)
* Progression Free Survival (PFS)
* Time to Progression (TTP)
* Time to next therapy

A total of 56 patients may be enrolled in this study: Dose escalation phase: Up to 24 subjects; Dose expansion phase: Up to a maximum of 38 patients treated at the maximum tolerated dose (MTD).

Study treatment will be administered starting at Cohort 1 for up to four sequential cohorts, with 3-6 patients in each cohort. A standard 3+ 3 dose escalation schedule will be used. A minimum of 3 patients will be entered within each cohort, to be expanded to 6 patients if dose limiting toxicities (DLTs) are observed, to determine the MTD. Once the MTD is reached, any additional patients will be enrolled at the MTD level.

Dose Escalation

* Cohort -1: bendamustine 120 mg/m2; pomalidomide 2mg; dexamethasone 40mg**
* Cohort 1 (initial dose): bendamustine 120/mg/m2; pomalidomide 3 mg; dexamethasone 40 mg**
* Cohort 2: bendamustine 120 mg/m2; pomalidomide 4 mg; dexamethasone 40 mg**
* Cohort 3: bendamustine 150 mg/m2; pomalidomide 4 mg; dexamethasone 40 mg**
* Cohort 4: bendamustine 180 mg/m2; pomalidomide 4 mg; dexamethasone 40 mg**

EVALUATION:

* For toxicity: 1 cycle (All patients will be considered evaluable for toxicity unless they cannot complete the first cycle of therapy due to withdrawal of consent or disease progression.)
* For efficacy: 2 cycles Intended treatment duration: Patients will continue on protocol as long as they are receiving clinical benefit and will be removed for disease progression (at the investigator's discretion the patient may be treated up to one cycle after progression noted to confirm progression), adverse event/unacceptable toxicity or side effect, or withdrawal of consent.

A DLT is defined as any of the following occurring during the first treatment cycle (28 days) that are judged by the investigator to be at least possibly related to the study therapy:

Hematologic:

* Febrile neutropenia (ANC <1.0x109/L) with fever of 38.5 C. Subjects who enter the study with lower counts (ANC <1.0x109/L) due to >5030%* marrow involvement will not be evaluated for this portion of the DLT definition.
* Grade 4 neutropenia (ANC < 0.5x109/L) for more than 7 days despite GCSF support. Subjects who enter the study with lower counts (ANC <1.0x109/L) due to >5030%* marrow involvement will not be evaluated for this portion of the DLT definition.
* Grade 4 thrombocytopenia (platelets count <25.0x109/L) lasting >7 days despite dose delay. Subjects who enter the study with lower counts (platelets <50.0x109/L) due to >5030%* marrow involvement will not be evaluated for this portion of the DLT definition.
* Grade 3-4 thrombocytopenia associated with bleeding
* Any hematologic toxicity requiring a dose reduction within Cycle 1
* Inability to receive Day 1 dose of Cycle 2 due to drug related toxicity persisting from Cycle 1 greater than 14 days

Non-hematologic:

* Any > Grade 3 toxicity determined by the Investigator to be related to pomalidomide or bendamustine (with the exception of thrombotic events and as noted below).
* > Grade 3 nausea, vomiting, or diarrhea, despite the use of maximal antiemetic/antidiarrheal therapy
* > Grade 3 neuropathy with pain
* >Grade 3 venous thromboembolic events.
* Any Grade 4 rash related to the agents will be considered a DLT.
* A Grade 3 rash related to the agents that has not resolved to < Grade 2 within a 10 day period despite steroids therapy will be considered a DLT.
* If an event is attributed to progressive disease, it will not be counted as a DLT.
* Any non-hematologic toxicity requiring a dose reduction within Cycle 1
* Delay in ability to receive Day 1 dose of Cycle 2 due to drug related toxicity persisting from Cycle 1 greater than 14 days

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all of the following inclusion criteria to be eligible to enroll in this study.

1. Cytopathologically or histologically confirmed diagnosis of multiple myeloma
2. Relapsed or refractory to most recent therapy (i.e. < 25% response, progression during therapy or within 60 days after completion).
3. Refractory to prior lenalidomide therapy (i.e. history of progression on therapy using full or maximally tolerated dose of lenalidomide for >/= two cycles).
4. Measurable disease:

   * Serum M protein > 0.5 g/dL or
   * Urine Bence Jones protein >200 mg/24 hr or
   * Elevated Free Light Chain per International Myeloma Working Group (IMWG) criteria, and abnormal ratio
5. Evidence of progression/relapse
6. Over 18
7. Life expectancy of more than 3 months
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
9. Total bilirubin < 2 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times ULN
10. Serum creatinine <3 mg/dL
11. • Absolute neutrophil count (ANC) >1.0 x 109/L or <1.0 x 109/L but > 0.75 due to >30%* marrow involvement (without granulocyte and granulocyte/macrophage colony stimulating factor (GCSF and GMCSF) for >1 week and of pegylated GCSF for >2 weeks)

    * Hemoglobin >8 g/dL
    * Platelet count >75.0 x 109/L or < 75.0 x 109/L but >50.0 x 109/L due to >30%* marrow involvement (without platelet transfusions for >1 week)
    * Transfusions allowed if clinically indicated
12. Agree to take enteric coated aspirin 81 mg daily
13. Consent
14. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test and abstain from sex or begin TWO acceptable methods of birth control >28 days before pomalidomide dose, and agree to ongoing pregnancy testing.
15. Male patients must abstain from sex or use a latex condom and not donate sperm while taking pomalidomide and for 1 week after stopping drug.
16. Register with POMALYST REMS™ and comply with their requirements.

EXCLUSION CRITERIA:

1. Patients with known sensitivity to immunomodulatory drugs (IMiDs)
2. Use of experimental drugs or therapy within 21 days of study-related drug therapy.
3. Exposure to chemotherapy or steroids within 14 days of study-related drug therapy.
4. Prior use of pomalidomide.
5. Radiation therapy within 14 days of screening.
6. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
7. Plasma cell leukemia.
8. Waldenström's macroglobulinemia.
9. Major surgery within 21 days prior to first dose.
10. Pregnant or lactating females.
11. Congestive heart failure, symptomatic ischemia, conduction abnormalities uncontrolled or myocardial infarction in the last six months.
12. Uncontrolled hypertension
13. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 14 days prior to first dose.
14. Active treatment or intervention for other malignancy or need active treatment within 8 months of starting study treatment.
15. Serious psychiatric or medical conditions that interfere with treatment
16. Significant neuropathy (Grade 3, Grade 4) at first dose and/or within 14 days before enrollment
17. Contraindication to required concomitant drugs
18. Patients with primary systemic amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2025-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gwynn Long, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2013. Dose escalation ended in November, 2013. Expansion enrollment began in December, 2013 and ended in September 2016. Patients were recruited from the Bone Marrow Transplant Clinic and Hematologic Malignancies Clinic at Duke University Medical Center.
Pre-assignment Details: Nine patients were consented to the study for cohort 1, however, 3 were screen failures. Seven patients were consented to the study for cohort 2, however, 5 were screen failures. Forty patients were consented to the study for the expansion phase, however, 10 were screen failures.
Groups:
- Cohort 1: 120mg Bendamustine + 3mg Pomalidomide; Cohort 2: 120mg Bendamustine + 4mg Pomalidomide: * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  After 6 cycles of treatment, dexamethasone may be decreased to 20mg. After total 12 cycles of treatment, subjects will proceed to the maintenance phase until time of progression.
  Study treatment will be administered starting at Cohort 1 for up to four sequential cohorts, with 3-6 patients in each cohort.
- Expansion: 120mg Bendamustine + 3mg Pomalidomide: * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  After 6 cycles of treatment, dexamethasone may be decreased to 20mg. After total 12 cycles of treatment, subjects will proceed to the maintenance phase until time of progression.
  Study treatment will be administered at the Maximum Tolerated Dose.
Period: Overall Study
Arm/Group | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide | Expansion: 120mg Bendamustine + 3mg Pomalidomide
Started | 6 | 2 | 30
Completed | 4 | 0 | 26
Not Completed | 2 | 2 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who received drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide | Expansion: 120mg Bendamustine + 3mg Pomalidomide | Total
Number analyzed (Participants) | 6 | 2 | 30 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 14 | 20
  >=65 years | 2 | 0 | 16 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 17 | 21
  Male | 4 | 0 | 13 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 29 | 37
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 5 | 6
  White | 6 | 1 | 25 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 30 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Pomalidomide and Bendamustine
Description: In the phase I dose escalation portion, patients will be sequentially enrolled in 4 cohorts at dose levels in a standard 3+3 design until the maximum tolerated dose (MTD) is reached.
  Cohort 1 (bendamustine 120mg/m2 + pomalidomide 3mg); Cohort 2 (bendamustine 120mg/m2 + pomalidomide 4mg); Cohort 3 (bendamustine 150mg/m2 + pomalidomide 4mg); Cohort 4 (bendamustine 180mg/m2 + pomalidomide 4mg)
  If dose limiting toxicity (DLT) is observed in 2 or more of the six patients at the same dosing level while DLT is observed in only 1 or none of the 6 patients at the dosing level immediately below it, then the lower dosing level will be defined as the maximum tolerated dose (MTD).
Time Frame: 2 cycles (approximately 2 months)
Population: All patients enrolled in cohort 1 and 2 evaluable for DLT. Cohorts 3 and 4 were not evaluated due to both patients in Cohort 2 experiencing DLT.
Measure: Number; unit: milligrams
Groups:
- Cohorts 1 and 2: * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
  Study treatment will be administered starting at Cohort 1 for up to four sequential cohorts, with 3-6 patients in each cohort. (Dose escalation)
  Bendamustine: Bendamustine 120mg/m2 (cohort 1, 2) or 150 mg/m2 (cohort 3), or 180mg/m2 (cohort 4) will be administered intravenously on day 1, every 28 days for 12 cycles.
  Pomalidomide: Pomalidomide 3mg (cohort 1) or 4mg (cohort 2, 3, 4) will be administered once daily orally (PO) on days 1-21, every 28 days until disease progression or death.
  Dexamethasone: Dexamethasone will be administered weekly orally or intravenously on days 1, 8,
Arm/Group | Cohorts 1 and 2
Number analyzed (Participants) | 8
milligrams
  Pomalidomide | 3
  Bendamustine | 120

2. Primary Outcome: Initial Response Rate
Description: The number of patients achieving a complete response (CR) or partial response (PR). Response is defined by the International Myeloma Working Group as:
  CR- Negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and < 5% plasma cells in bone marrow
  PR- > 50% reduction of serum M-protein and urine M-protein by >90% or to < 200 mg/24 h In addition, if present at baseline, a > 50% reduction in the size of soft tissue plasmacytomas is also required
  VGPR - Serum and urine M-protein detectable by immunofixation but n
Time Frame: 2 cycles (approximately 2 months)
Population: The overall number of participants analyzed reflects those who received at least 2 cycles of treatment. These participants were assessed for response at that time. The data reported indicates how many patients out of each cohort experienced at least a partial response or complete response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide | Expansion: 120mg Bendamustine + 3mg Pomalidomide
Number analyzed (Participants) | 5 | 0 | 27
Participants
  Partial Response | 1 |  | 11
  Very Good Partial Response | 0 |  | 2
  Complete Response | 0 |  | 0

3. Secondary Outcome: Overall Response Rate
Description: The number of patients achieving stable disease (SD), partial response (PR), very good partial response (VGPR), complete response (CR) or stringent complete response (sCR)
  sCR = CR as defined in Primary Outcome measure 2 plus normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  VGPR = Serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h
  SD = Not meeting criteria for CR, VGPR, PR, or progressive disease
Time Frame: 2 years after last dose of study drug
Reporting Status: Not Posted

4. Secondary Outcome: Time to Progression
Description: Time to progression - defined as time elapsed in patients between achievement of response and disease progression
Time Frame: 2 years after last dose of study drug
Reporting Status: Not Posted

5. Secondary Outcome: Time to Next Therapy
Description: Time to next Therapy - defined as the time elapsed for patients from initiation of study therapy until initiation of next therapy
Time Frame: 2 years after last dose of study drug
Reporting Status: Not Posted

6. Secondary Outcome: Progression Free Survival
Description: The time elapsed for patients between initiation of study therapy and either disease progression or death
Time Frame: 2 years after last dose of study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days past last day of drug, up to 1 year
Description: Adverse Events were not collected per cohort, so they are represented as a whole
Groups:
- Cohort 1: 120mg Bendamustine + 3mg Pomalidomide; Cohort 2: 120mg Bendamustine + 4mg Pomalidomide; Expansion: 120mg Bendamustine + 3mg Pomalidomide: * Pomalidomide: once daily oral (PO) dosing on days 1-21, every 28 days
  * Bendamustine: once intravenous (IV) dosing on day 1, every 28 days
  * Dexamethasone: weekly PO or IV dosing on days 1, 8, 15, and 22 every 28 days
Arm/Group | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide | Expansion: 120mg Bendamustine + 3mg Pomalidomide
All-Cause Mortality (participants affected / at risk) | 6/6 | 2/2 | 13/30
Serious Adverse Events (participants affected / at risk) | 6/6 | 1/2 | 17/30
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide (N=6) | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide (N=2) | Expansion: 120mg Bendamustine + 3mg Pomalidomide (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1) | 9 (9)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 4 (5) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 120mg Bendamustine + 3mg Pomalidomide (N=6) | Cohort 2: 120mg Bendamustine + 4mg Pomalidomide (N=2) | Expansion: 120mg Bendamustine + 3mg Pomalidomide (N=30)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 23 (73)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 5 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 11 (17)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 1 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 21 (46)
Fever (General disorders) | 1 (5) | 1 (1) | 4 (7)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 3 (7)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 8 (13)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 3 (8)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 10 (22)
Neutrophil count decreased (Investigations) | 4 (9) | 1 (1) | 26 (53)
Platelet count decreased (Investigations) | 3 (6) | 1 (1) | 20 (41)
Weight loss (Investigations) | 0 (0) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 19 (36)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 10 (23)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 15 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 15 (29)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 14 (30)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 18 (32)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 8 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (11)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 11 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (9)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 11 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 5 (7)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 14 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 15 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (11)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes